CLINICAL TRIAL: NCT05228886
Title: Intensifying Community Referrals for Health: The SINCERE Intervention to Address COVID-19 Health Disparities
Brief Title: The SINCERE Intervention to Address COVID-19 Health Disparities
Acronym: SINCERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Wallace (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Andrea Wallace, Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00140301; 1R01NR019944-01 (NIH)
Record Dates: First submitted 2022-02-03; First posted 2022-02-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Vulnerable Populations; Social Determinants of Health
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Services to which participants are referred will not be aware of the participant's inclusion in the research study or their study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Call + Resources (Active Comparator): Participants receive standard care typically provided to 211 callers, including ad hoc follow-up.
  Interventions: Other: Standard of Care
- Call + Resources + Scheduled Follow-Up (Experimental): Participants receive standard care typically provided to 211 callers plus scheduled follow-up calls according to the Scheduled Follow-Up intervention description.
  Interventions: Behavioral: Scheduled Follow-Up
- Call + Resources + SINCERE (Experimental): Participants receive standard care typically provided to 211 callers plus scheduled follow-up calls according to the SINCERE intervention description (scheduled follow up with active collaborative goal setting).
  Interventions: Behavioral: SINCERE

INTERVENTIONS:
Behavioral: SINCERE — Each goal setting session will involve templated prompts in 211's ServicePoint to guide the creation of a patient-centered "action plan" specifying what, when, how much, and how often patients will engage in a behavior (e.g., "I will work on filling out eligibility paperwork for 30 minutes on Wednesday evening"). Again, following clear prompts, ISs negotiate the "action plan" with patients until patients can rate their level of confidence for achieving this behavior a 7 on a scale from 0 to 10.
  Arms: Call + Resources + SINCERE
Behavioral: Scheduled Follow-Up — Adding to the standard Call + Resources protocol, those assigned to scheduled follow-up will receive a proactive call from 211 every 2 weeks for 3 months to explore additional service needs. These calls will be unstructured, guided by participant requests and 211 IS prompts.
  Arms: Call + Resources + Scheduled Follow-Up
Other: Standard of Care — 211 ISs contact referred patients, provide referral services, and follow up in an ad-hoc manner.
  Arms: Call + Resources

SUMMARY:
The goal of this real world efficacy study is to understand the benefit of universal social needs screening, community-based service referrals, and telephonic follow-up as a scalable strategy for preventing COVID-19 transmission, and for addressing the secondary health effects of the social, behavioral, and economic changes following the COVID-19 pandemic. With statewide community service providers, existing health information technology, and piloted methods, we seek to determine the effectiveness of universal social needs screening and community service referrals - the SINCERE intervention - in improving health outcomes of COVID-19 vulnerable and socioeconomically disadvantaged populations and whether intensive follow-up and collaborative goal-setting helps overcome barriers to community service use by patients seen in the emergency department and seeking COVID testing at community-based and mobile clinic locations.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 17 years)
* English or Spanish speaking
* Completed the referral process at the UHealth ED, one of the COVID-19 testing sites or the Primary Children's ED and indicated both social needs and willingness to receive service low- and no-cost referrals from the United Way 211 community referral service
* Able to be reached by phone during the intervention OR able to complete surveys sent by text or email

Exclusion Criteria:

* Those unable to communicate verbally
* Those living in nursing facilities, or those who are not otherwise responsible for self-care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Global Health over 12-week time period | Baseline, 2-week, 4-week and 12-week surveys
  Standardized PROMIS v1.2 Global Health. 10 questions create one outcome score. Each question is on a 1-5 scale with higher numbers indicating lower severity. The outcome variable will be PROMIS v1.2 Global Health with Time included as a variable in the model.
Change in Depression over 12-week time period | Baseline, 2-week, 4-week and 12-week surveys
  Standardized PROMIS Depression - Short Form 8b. 8 questions create one outcome score. Each question is on a 1-5 scale with higher numbers indicating higher severity. The outcome variable will be PROMIS Anxiety with Time included as a variable in the model.
Change in Anxiety over 12-week time period | Baseline, 2-week, 4-week and 12-week surveys
  Standardized PROMIS Anxiety- Short Form 7a. 7 questions create one outcome score. Each question is on a 1-5 scale with higher numbers indicating higher severity. The outcome variable will be PROMIS Anxiety with Time included as a variable in the model.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wallace, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
In agreement with the investigative team, the PI will share de-identified data to other investigators for study. Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and can be used for secondary study purposes. The PI agrees to make available data within one year of the completion of the funded project period and manuscripts pertaining to the Aims. De-identified data will be available directly from the PI after consulting with the investigative team on relevant requests. The PI agrees to share data in a manner that is fully consistent with NIH data sharing policies and applicable laws and regulations.